CLINICAL TRIAL: NCT03705624
Title: P. Falciparum Infection Dynamics and Transmission to Inform Elimination (INDIE-1a)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre national de recherche et de formation sur le paludisme (Other Government); Radboud University Medical Center (Other); Institute for Disease Modeling, Bellevue, US (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INDIE-1a
Record Dates: First submitted 2018-07-19; First posted 2018-10-15 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2018-08

CONDITIONS: Malaria
Keywords: falciparum; gametocyte; elimination; anopheles; transmission; diagnostic
MeSH Terms: conditions — Malaria; Disease | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Standard of care with passively monitored malaria incidence at health centers that receive appropriate diagnostic and clinical supplies and Seasonal Malaria Chemoprevention (SMC) for children less than 5 years of age
- CCM (Experimental): Standard of care supplemented with enhanced Community Case Management for malaria (CCM) involving weekly active screening for fever using a research-grade thermometer by a trained health worker. A measured temperature ≥37.5°C or reported fever in the last 24 hours will prompt screening with a conventional rapid diagnostic test (RDT). RDT positive individuals will be treated with artemether-lumefantrine (AL) according to national guidelines
  Interventions: Other: Enhanced Community Case Management (CCM)
- CCM+MSAT (Experimental): Standard of Care supplemented with CCM and Monthly Screening and Treatment (MSAT) regardless of symptoms with a conventional RDT. Screening will be performed by research staff with 25-35 days between screening rounds; RDT positive individuals will be treated with AL according to national guidelines.
  Interventions: Other: Enhanced Community Case Management (CCM); Other: Monthly Screening and Treatment (MSAT)

INTERVENTIONS:
Other: Enhanced Community Case Management (CCM) — Enhanced Community Case Management for malaria (CCM) involving weekly active screening for fever using a research-grade thermometer by a trained health worker. A measured temperature ≥37.5°C or reported fever in the last 24 hours will prompt screening with a conventional rapid diagnostic test (RDT). RDT positive individuals will be treated with AL according to national guidelines
  Arms: CCM; CCM+MSAT
Other: Monthly Screening and Treatment (MSAT) — Monthly Screening and Treatment (MSAT) regardless of symptoms with a conventional RDT. Screening will be performed by research staff with 25-35 days between screening rounds; RDT positive individuals will be treated with AL according to national guidelines.
  Arms: CCM+MSAT

SUMMARY:
In the current randomized trial, the investigators will test the ability of two experimental approaches to malaria infection management to reduce malaria transmission potential. Compounds in Saponé, Burkina Faso, will be randomized to 1 of 3 study arms: arm 1 - current standard of care with passively monitored malaria infections; arm 2 - standard of care plus enhanced community case management (CCM), comprising active weekly screening for fever, and detection and treatment of infections in fever positive individuals using conventional rapid diagnostic tests (RDTs); or arm 3 - standard of care and enhanced CCM, plus monthly screening and treatment (MSAT) using RDTs. The study will be conducted over approximately 18 months covering two high transmission seasons and the intervening dry season

ELIGIBILITY:
Inclusion Criteria:

1. Participants should be permanent residents of the compound
2. Participants should be willing to participate in repeated assessments of health and infection status and willing to donate a maximum of 37mL of blood (children <10 years of age) or 52mL of blood (older individuals) during an 18-month period

Exclusion Criteria:

1. Any (chronic) illness that would affect with study participation
2. Pre-existing severe chronic health conditions
3. Current participation in malaria vaccine trials or participation in such trials in the last 2 years
4. History of intolerance to artemether-lumefantrine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Parasite prevalence and density by molecular detection at the end of study cross-sectional survey. | Month 18 (end of second transmission season; January-February 2020)
  The primary outcome measure is parasite prevalence in the cross-sectional survey conducted at the end of the transmission season of year 2. If CCM and MSAT result in the early detection of infections, parasite prevalence at the end of the study will be lower in these arms compared to the control arm.

SECONDARY OUTCOMES:
Parasite prevalence and density by molecular detection at the end of year 1 cross-sectional survey. | Month 6 (end of first transmission season; January-February 2019)
  Parasite prevalence and density in the cross-sectional survey conducted at the end of the transmission season of year 1. If CCM and MSAT result in the early detection of infections, parasite prevalence will be lower in these arms compared to the control arm.
Parasite prevalence and density by molecular detection at the end of dry season cross-sectional survey. | Month 12 (prior to second transmission season; June 2019)
  Parasite prevalence and density in the cross-sectional survey conducted at the end of the dry season. If CCM and MSAT result in the early detection of infections, parasite prevalence will be lower in these arms compared to the control arm.
Gametocyte prevalence and or density in P. falciparum infections at the end of study cross-sectional survey | Month 18 (end of second transmission season; January-February 2020)
  Gametocyte prevalence in qPCR detected infections is assessed by molecular methods and compared between study arms.
Gametocyte prevalence and or density in P. falciparum infections at the end of year 1 cross-sectional survey | Month 6 (end of first transmission season; January-February 2019)
  Gametocyte density of male and female gametocytes will be assessed by molecular methods and compared between study arms.
Gametocyte prevalence and or density in P. falciparum infections at the end of dry season cross-sectional survey | Month 12 (prior to second transmission season; June 2019)
  Gametocyte density of male and female gametocytes will be assessed by molecular methods and compared between study arms.
Gametocyte prevalence and or density in P. falciparum during all study visits | Throughout study, an average of 18 months
  Gametocyte density of male and female gametocytes will be assessed by molecular methods and compared between study arms.
The number of incident infections. | Throughout study, an average of 18 months
  Regular visits by CCM and MSAT will result in the identification of malaria infections that are not detected during passive case detection. The numbers of infections that are detected in each arm are quantified and compared between arms.
Infectivity to mosquitoes of P. falciparum infections | Throughout study, an average of 18 months
  For a selection of infections, infectiousness to mosquitoes is assessed by membrane feeding assays.

OTHER OUTCOMES:
The detectability of infections by highly sensitive rapid diagnostic tests. | Throughout study, an average of 18 months
  For a selection of samples, the detectability of infections is assessed by conventional rapid diagnostic test and by highly sensitive rapid diagnostic tests and related to i. histidine rich protein-2 (HRP2) concentrations; ii. duration of infection; iii. parasite density by molecular diagnostics.
The relationship between the proportion of infected mosquitoes and gametocyte density. | Throughout study, an average of 18 months.
  Gametocyte density and sex ratio will be assessed by molecular methods and associated with the proportion of infected mosquitoes and the burden of infection in mosquitoes
The impact of infection characteristics on the transmissibility of infections to mosquitoes | Throughout study, an average of 18 months.
  Under this outcome, we aim to determine the impact of gametocyte sex-ratio, other gametocyte characteristics, duration of infection and clonal complexity of malaria infections on the transmissibility of infections to mosquitoes
The impact of human host characteristics on the transmissibility of infections to mosquitoes | Throughout study, an average of 18 months
  Under this outcome, we aim to determine the impact of red blood cell haemoglobinopathies, haemoglobin concentration, inflammatory markers, naturally acquired antibody responses to gametocyte antigens and other host characteristics on the transmissibility of infections to mosquitoes
Association between total parasite density and gametocyte density | Throughout study, an average of 18 months
  Under this outcome, we aim to evaluate the relationship between asexual parasite density and gametocyte density in P. falciparum infections
Malaria transmission potential based on measured gametocyte densities | Throughout study, an average of 18 months
  Under this outcome, we aim to determine malaria transmission potential of infections based on the gametocyte density
Number of acquired clones based on genotyping | Throughout study, an average of 18 months
  Under this outcome, we aim to examine the complexity of P. falciparum infection by measuring the number of clones present in infections
The duration of infections in the dry season | Month 6-12, between end of season survey January/February 2019 and end of dry season survey June 2019
  Under this outcome, we aim to evaluate the duration of P. falciparum carriage during the dry season
To quantify mosquito exposure in relation to incident infections | Throughout study, an average of 18 months
  Under this outcome, we aim to quantify mosquito exposure and relate this to number of incident infections

CONTACTS AND LOCATIONS:
Overall Officials: Chris Drakeley, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine, Faculty of Infectious and Tropical Diseases, London, United Kingdom; Alfred Tiono, PhD, MD, Principal Investigator — Centre national de recherche et de formation sur le paludisme; Teun Bousema, PhD, Principal Investigator — Radboud university medical centre, Nijmegen, The Netherlands
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual participant data may be shared on a digital repository or upon reasonable request.

REFERENCES:
- [Derived] Collins KA, Ouedraogo A, Guelbeogo WM, Soulama I, Ouattara MS, Sombie S, Ouedraogo N, Coulibaly AS, Nombre A, Lanke K, Ramjith J, Awandu SS, Serme SS, Henry N, Stone W, Ouedraogo IN, Diarra A, Holden TM, Sirima SB, Bradley J, Soremekun S, Selvaraj P, Gerardin J, Drakeley C, Bousema T, Tiono AB. Effect of weekly fever-screening and treatment and monthly RDT testing and treatment on the infectious reservoir of malaria parasites in Burkina Faso: a cluster-randomised trial. Lancet Microbe. 2024 Sep;5(9):100891. doi: 10.1016/S2666-5247(24)00114-9. Epub 2024 Jul 25. PMID 39068937
- [Derived] Collins KA, Ouedraogo A, Guelbeogo WM, Awandu SS, Stone W, Soulama I, Ouattara MS, Nombre A, Diarra A, Bradley J, Selvaraj P, Gerardin J, Drakeley C, Bousema T, Tiono A. Investigating the impact of enhanced community case management and monthly screening and treatment on the transmissibility of malaria infections in Burkina Faso: study protocol for a cluster-randomised trial. BMJ Open. 2019 Sep 13;9(9):e030598. doi: 10.1136/bmjopen-2019-030598. PMID 31519680